CLINICAL TRIAL: NCT02928159
Title: Low Pulse Amplitude Seizure Therapy (LAP-ST Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Behman Hospital (Other)
Responsible Party: Principal Investigator, Emad Sidhom, Physician, Behman Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 001
Record Dates: First submitted 2016-10-05; First posted 2016-10-10 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Mood Disorders; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Low Pulse Amplitude Seizure Therapy; Electroconvulsive Therapy; Low Pulse Amplitude Electroconvulsive Therapy; Low Pulse Amplitude ECT; LAP; LAP-ST; ECT; Mood disorders; Psychotic disorders
MeSH Terms: conditions — Mood Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Pulse Amplitude Seizure Therapy (Experimental): Course of Right Unilateral Ultrabrief LAP-ST using Mecta spectrum 5000Q Device.
  Interventions: Device: Mecta spectrum 5000Q device

INTERVENTIONS:
Device: Mecta spectrum 5000Q device — LAP-ST and Right Unilateral (RUL) electrode placement.

SUMMARY:
This study assesses the feasibility of a full course of Low Pulse Amplitude-Seizure Therapy (LAP-ST) (primary outcome).

DETAILED DESCRIPTION:
This is hypothesized to increase stimulation focality, thus minimizing cognitive side effects compared to conventional ECT. The study will enroll 22 patients recruited from the Behman Hospital, Cairo, Egypt. Patients referred to ECT service in the Behman Hospital who are clinically indicated to do ECT for major depressive episode of a mood disorder or psychotic episode of a primary psychotic disorder will be approached. Eligible participants who signed informed consent will be included to receive a course of Right Unilateral Ultrabrief LAP-ST.

ELIGIBILITY:
Inclusion Criteria:

1. ECT clinically indicated
2. Males or females over 22 to 80 years of age
3. Use of effective method of birth control for women of child-bearing capacity
4. Patient is medically stable
5. Capacity of patient to fully participate in the informed consent process as evaluated by their clinician

Exclusion Criteria:

1. Current unstable or serious medical condition, or any co-morbid medical condition that substantially increases the risks of ECT
2. History of conditions that may make ECT unsafe such as metal in the head, or a skull defect
3. Female patients who are currently pregnant or plan to be pregnant during the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Feasibility (by successfully inducing therapeutic seizures during LAP-ST course) | From first to last session of LAP-ST course (average approximately 2 weeks)
  Measured by: the elicitation of therapeutic seizure in the brain and assessed by using EEG

SECONDARY OUTCOMES:
Memory (cognitive side effects) | From Baseline to end of acute course (average 2 weeks)
  Measured by: Mini Mental State Examination
Time to reorientation | From Baseline to end of acute course (average 2 weeks)
  Measured by: Time to Orientation Test
Efficacy | From Baseline to end of acute course (average 2 weeks)
  Montgomery-Åsberg Depression Rating Scale (MADRS) for depressive episodes of mood disorders
Efficacy | From Baseline to end of acute course (average 2 weeks)
  Brief Psychiatric Rating Scale (BPRS) for psychotic disorders

CONTACTS AND LOCATIONS:
Overall Officials: Nagy A. Youssef, Principal Investigator — Medical College of Georgia, Augusta University; Emad Sidhom, Principal Investigator — Behman Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Youssef NA, Sidhom E. Feasibility, safety, and preliminary efficacy of Low Amplitude Seizure Therapy (LAP-ST): A proof of concept clinical trial in man. J Affect Disord. 2017 Nov;222:1-6. doi: 10.1016/j.jad.2017.06.022. Epub 2017 Jun 16. PMID 28667887